CLINICAL TRIAL: NCT05718895
Title: An Open, Multi-center, Phase I Clinical Study of ATG 022 in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Study of ATG-022 in Patients With Advanced/Metastatic Solid Tumors
Acronym: CLINCH
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Antengene Biologics Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATG-022-ST-001
Record Dates: First submitted 2023-01-17; First posted 2023-02-08 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Intervention Model Description: A treatment cycle of ATG-022 will be defined as 21 days. Dosing will begin at 0.3 mg/kg Q3W with 1 subject
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-022 (Experimental): Dose Escalation Phase:
  for subjects with solid tumors,approximately 16-36 subjects will be enrolled .
  Dose Expansion Phase:
  The tumor types in the Dose Expansion Phase may involve other tumor types based on the signals from the Dose Escalation Phase. The total number of patients in dose expansion will be up to approximately 120 patients.
  Interventions: Drug: ATG-022

INTERVENTIONS:
Drug: ATG-022 — Dose Escalation Phase:
  A treatment cycle of ATG-022 will be defined as 21 days. Dosing will begin at 0.3 mg/kg once every 3 weeks (Q3W) with 1 subject ,the following dose cohorts (0.9, 1.8, 2.4, 3.0, and 3.6 mg/kg Q3W) will require at least 3 and up to 6 evaluable subjects by using dose escalation plan of "3+3" design.

SUMMARY:
This is an Open, Multi-center, Phase I Clinical Study of ATG 022 in Patients with Advanced/metastatic Solid Tumors

DETAILED DESCRIPTION:
This is a Phase I, multi-center, open-label, dose-finding study of ATG-022 in patients with advanced solid tumours. The study design includes a Dose Escalation Phase which will enroll subjects with advanced/metastatic solid tumors, and a Dose Expansion Phase which will enroll select advanced/metastatic solid tumors with Claudin 18.2-positive expression at the defined maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) to further evaluate the safety, tolerability, and efficacy of ATG-022.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures, sampling, and analyses.
2. Aged at least 18 years as of the date of consent.
3. Histological or cytological confirmation of a solid tumor, and have progressed despite standard therapy(ies), or are intolerant to standard therapy(ies), or not applicable for standard therapy(ies).

   1. Dose Escalation Phase: all solid tumors.
   2. Dose Expansion Phase: Claudin 18.2 positive solid tumors.
4. Subjects should be willing to receive a biopsy at screening, if no former available tumor tissue samples within 36 months prior to participating in the study are provided.
5. At least 1 measurable lesion per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
6. Estimated life expectancy of a minimum of 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 .
8. Females should be using adequate contraceptive measures until 180 days after the end of treatment, should not be breastfeeding, and must have a negative pregnancy test prior to the start of dosing if of child-bearing potential or must have evidence of nonchild-bearing potential by fulfilling one of the following criteria at screening
9. Male subjects should be willing to use effective contraception, ie condoms, for the duration of the study and 180 days after the final dose of study treatment.

Exclusion Criteria:

1. Primary central nervous system disease or central nervous system metastatic disease.
2. Prior exposure to a Claudin 18.2 targeting agent.
3. Prior therapy with any chemotherapy, immunotherapy, anticancer agents, or investigational products from a previous clinical study within 28 days of the first dose of study treatment or within a period during which the investigational product or systemic anticancer treatment has not been cleared from the body (eg, a period of 5 'half-lives'.
4. Prior vaccination within 28 days of the first dose of study therapy.
5. Prior any solid organ transplant. Autologous stem cell transplant or CAR-T cell infusion < 6 months prior to the first dose of study treatment.
6. Active infection including hepatitis B, and/or hepatitis C.
7. Known history of human immunodeficiency virus (HIV) infection.
8. Any unresolved toxicities from prior therapy greater than Grade 1 at the time of ICF signature, with the exception of alopecia.
9. Pregnant or nursing females.
10. History of hypersensitivity or history of allergic reactions attributed to drugs with a similar chemical or biologic structure or class to ATG-022.
11. Other primary malignancies developed within 5 years prior to the first dose of the study drug, except locally curable malignancies after radical treatment .
12. In the opinion of the investigator, subject's complications, or other conditions (psychological, familial, sociological, or geographical etc.) may affect protocol compliance or may be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 21 Days
  Number of Participants with Dose Limiting Toxicity
MTD | Up to 21 Days
  Maximum Tolerated Dose
RP2D | Up to 21 Days
  RP2D= Recommended Phase 2 Dose

SECONDARY OUTCOMES:
PFS | 12 months after the last subject enrolled
  Progression Free Survival
ORR | 12 months after the last subject enrolled
  Overall Response Rate
DOR | 12 months after the last subject enrolled
  Duration of Response

OTHER OUTCOMES:
OS | 12 months after the last subject enrolled
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (16):
- Australia (3):
  - Cancer Research SA Pty Ltd, Adelaide
  - Cabrini Health Limited, Malvern
  - Integrated Clinical Oncology Network Pty Ltd (Icon), South Brisbane
- China (13):
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Jinan Central Hospital, Jinan
  - Gansu provincial cancer hospital [recruiting], Lanzhou
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tongren Hospital Shanghai, Shanghai
  - Liaoning Cancer Hospital, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiangzhuang
  - Shanxi provincial cancer hospital, Taiyuan
  - Hubei Cancer Hospital, Wuhan
  - The First affiliated hospital of Xi'An Jiao Tong Ubiversity, Xi'an
  - Xuzhou Central Hospital, Xuzhou